CLINICAL TRIAL: NCT01469507
Title: Comparative Study of Efficacy and Safety of Three Intra Articular Injections of V0220 Versus Hyalgan® in Patients Suffering From Symptomatic Knee Osteoarthritis. A Multinational Multicentric, Randomised, Double-blind, Parallel-group Study
Brief Title: Efficacy and Safety Study in Patients Suffering From Knee Osteoarthritis
Acronym: VESTA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V00220 IA 0 01; 2011-002295-17 (EudraCT Number)
Record Dates: First submitted 2011-11-07; First posted 2011-11-10 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- V0220 (Experimental)
  Interventions: Device: Chondroitin sulfate and sodium hyaluronate
- Hyaluronan (Active Comparator)
  Interventions: Drug: Hyaluronan

INTERVENTIONS:
Device: Chondroitin sulfate and sodium hyaluronate — 3 weekly injections
  Arms: V0220
Drug: Hyaluronan — 3 weekly injections
  Other Names: Hyalgan®
  Arms: Hyaluronan

SUMMARY:
The primary objective of this study is to compare a combination of hyaluronic acid and chondroitin sulfate (V0220) to Hyalgan® on pain relief in patients with symptomatic knee osteoarthritis (OA) over 24 weeks when administered in three weekly injections.

Chondroitin sulfate is one of the components of cartilage. Studies have shown that chondroitin sulphate improves the quality of the hyaluronic acid produced in the joint. The benefit of V0220 combination is based on two main physicochemical properties, in line with the characteristics of osteoarthritic disease: optimising the rheological behaviour and improving the buffering effect on synovial flow ("outflow buffering").

ELIGIBILITY:
Inclusion Criteria:

* presenting with uni or bilateral medial and/or lateral femorotibial osteoarthritis of the knee evolving for more than 6 months
* patients taking analgesic medications for at least 3 months prior to randomisation and dissatisfied with their current therapy

Exclusion Criteria:

* isolated symptomatic femoropatellar osteoarthritis
* target knee prothesis
* having undergone an articular lavage, or an arthroscopy or any surgery on the target knee in the 6 months preceding randomisation,
* target knee osteoarthritis with clinical joint effusion at selection and at randomization
* body mass index (BMI) greater than or equal to 30,
* patient having received any corticosteroid treatment by any administration route (other than inhalers, ocular, auricular route) in the month preceding randomisation,
* patient having received intra-articular steroid injection in the target knee within the month preceding randomisation or patient having received intra-articular hyaluronic acid in the target knee in the 6 months preceding randomisation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Pain relief assessed on a global pain Visual Analogic Scale | change from baseline over 24 weeks

SECONDARY OUTCOMES:
Functional improvement (questionnaire) | change from baseline over 24 weeks
Patient's and investigator's global assessment of the disease status (Visual Analogic Scale ) | change from baseline over 24 weeks
Patient's health related quality of life (questionnaire) | over 24 weeks
Consumption of analgesic medication (paracetamol and NSAIDs)(number of days and quantity) | over 24 weeks
Medico-economic questionnaire | over 24 weeks
Occurrence of adverse events | over 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel MAHEU, Dr, Principal Investigator — private practice / unaffiliated